CLINICAL TRIAL: NCT04513223
Title: Safety, Tolerability, Pharmacokinetics, and Antitumour Activity of SHR-A1811, in Patients With HER2-expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma and Colorectal Cancer: a Phase 1 Study
Brief Title: A Phase 1 Study of SHR-A1811 in Patients With Selected HER2 Expressing Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-I-102
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — There are six pre-defined dose regimens . Subjects will be enrolled with an initial dose

SUMMARY:
This is a single arm, open-label, dose escalation, PK expansion and efficacy expansion study of phase I. The purpose of this study is to assess the tolerability, safety, pharmacokinetics and immunogenicity of SHR-A1811 and preliminary anti-tumor efficacy in HER2-expressing advanced gastric or gastroesophageal junction adenocarcinoma and colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically or cytologically documented advanced/unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma and colorectal cancer that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* At least one evaluable or measurable lesion should be present and identified according to Response Evaluation Criteria in Solid Tumors(RECIST) version 1.1.
* Has an ECOG PS 0-1.
* Has a life expectancy of ≥ 3 months.
* Has adequate organ function

Exclusion Criteria:

* Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0 grade ≤ 1.
* Has received HER2 antibody drug conjugates,.
* Central nervous system metastasis or meningeal metastasis with clinical symptoms
* Has active infection requiring systemic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
DLT and the recommended Phase 2 dose (RP2D) | Subjects will be treated and observed for dose-limiting toxicity(DLT) through the end of the first cycle (Days 1-21).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided